CLINICAL TRIAL: NCT06033859
Title: Incidence of Bleeding on Probing as an Indicator of Peri-Implant Disease Progression: A Prospective Study
Brief Title: Incidence of Bleeding on Probing as an Indicator of Peri-Implant Disease Progression
Acronym: BOP
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Andrea Ravida, Assistant Professor, University of Pittsburgh
Other Study IDs: STUDY22060166
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Peri-Implantitis; Bleeding of Subgingival Space
Keywords: Bleeding on probing; Peri-implant mucositis
MeSH Terms: conditions — Peri-Implantitis | interventions — Dental Prophylaxis; Maintenance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Implants with BOP score 0: Implants with no BOP according to the modified bleeding index at baseline.
  Interventions: Diagnostic Test: Clinical measurements; Diagnostic Test: Radiographic measurement; Procedure: Dental prophylaxis or maintenance
- Implants with BOP score 1: Implants with a bleeding dot at baseline.
  Interventions: Diagnostic Test: Clinical measurements; Diagnostic Test: Radiographic measurement; Procedure: Dental prophylaxis or maintenance
- Implants with BOP score 2: Implants with a continuous line of blood that fills the sulcus at baseline.
  Interventions: Diagnostic Test: Clinical measurements; Diagnostic Test: Radiographic measurement; Procedure: Dental prophylaxis or maintenance
- Implants with BOP score 3: Implants with a profuse bleeding and/or hemorrhage drip at baseline.
  Interventions: Diagnostic Test: Clinical measurements; Diagnostic Test: Radiographic measurement; Procedure: Dental prophylaxis or maintenance

INTERVENTIONS:
Diagnostic Test: Clinical measurements — With the aid of a periodontal probe, the incidence of BOP, as well as PD, recession and KM will be assessed.
Diagnostic Test: Radiographic measurement — A standardized periapical radiograph of the implant will be completed at the beginning and the end of study to determine the marginal bone loss.
Procedure: Dental prophylaxis or maintenance — Dental prophylaxis or maintenance will be performed every 3 months.

SUMMARY:
The primary goal of the present prospective cohort study is to evaluate the effect of varying incidences of BOP at implant sites across 15 months of maintenance visits on the probability of peri-implant disease progression. Over 15 months, participants will attend 6 visits where clinical measurements and maintenance care will be performed every 3 months.

DETAILED DESCRIPTION:
Screening/Baseline/Maintenance Visit 1 (V1) After participants have consented, their health history will be reviewed, and their vitals including blood pressure and heart rate will be recorded. A dental exam of the teeth and gums will be completed. During this exam, a UNC 15 periodontal probe will be used to perform the clinical assessments. Intraoral photographs will be taken. An x-ray of the implant(s) included in the study will be taken using a customized x-ray holder (created during Visit 1) so that at the end of the study, a final x-ray will be taken in the exact same position. Finally, each participant will receive a dental prophylaxis (D1110) or maintenance (D4910) according to their prior periodontal diagnosis.

Maintenance Visits 2-6 (V2-V6) Participants will return in 3-month intervals at approximately 3, 6, 9, 12, and 15 months (+/- 10 days) for Study Visits V2 - V6. At each of these visits, individuals will be asked about continued participation in the study. Participants will also be asked if there have been any changes to medical or dental history and if they are taking any new medications. Intraoral photographs of the study area will be performed, as well as, collecting measurements from around the dental implant(s), and providing regular dental cleaning. At the 15 month visit, a final x-ray will be taken using the custom x-ray holder made at the first visit.

Clinical and radiographic assessments will include:

1. BOP: at each of the 4 measured locations surrounding the implant of interest will be recorded as follows:

   1. Score 0 - No BOP
   2. Score 1 - Bleeding dot
   3. Score 2 - Continuous line of blood that fills the sulcus
   4. Score 3 - Profuse bleeding and/or hemorrhage drip.
2. Probing depths (PD): at 4 locations surrounding the implant of interest (mesiolingual (ML), mesiobuccal (MB), distolingual (DL), and distobuccal (DB)). PD increase must exceed a threshold of 0.8mm to be considered progression.
3. Recession: measured at each of the 4 locations surrounding the implant of interest.
4. Keratinized mucosa width: measured at the midbuccal aspect of the implant(s).
5. Mucosal thickness: assessed with the aid of an endodontic spreader, 2mm below the mucosal margin, at the midbuccal aspect of the implant(s).
6. Marginal bone loss (MBL): measured by overlaying the baseline and final radiographs and measuring the change in marginal bone levels. Progression will have to exceed a threshold of 0.5mm to be considered.

ELIGIBILITY:
Inclusion Criteria:

To be enrolled in the study, the participant must meet the following inclusion criteria:

* adults in good general health (at least ASA 2)
* having ≥ 1 dental implant that was restored before January 2021
* patients of the University of Pittsburgh Periodontics Department
* available for maintenance visits every 3 months for the length of the study

Exclusion Criteria:

* Active infectious diseases of any kind
* Pregnant or planning to become pregnant (self-reported)
* Congenital or metabolic bone disorders
* Current heavy smokers: Subjects who have smoked more than 1 pack/day within 6 months of study onset
* Co-morbid conditions that would affect the study outcome or interpretation of study results
* Require treatment for periodontal disease prior to baseline

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population from which cases will be recruited are from the patients of record at the University of Pittsburgh Periodontics Department who meet the inclusion criteria of the study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Marginal Bone Loss (MBL) | Baseline and 15 months
  MBL will be calculated by measuring the difference in marginal bone level between the standardized periapical radiographs. Progression will have to exceed a threshold of 0.5mm to be considered.

SECONDARY OUTCOMES:
Incidence of BOP | 3, 6, 9, 12 and 15 months
  Changes in BOP at each of the 4 sites assessed in baseline, according to Mombelli et al. (1987):
  1. Score 0 - No BOP
  2. Score 1 - Bleeding dot
  3. Score 2 - Continuous line of blood that fills the sulcus
  4. Score 3 - Profuse bleeding and/or hemorrhage drip.
Changes in probing depth (PD) | Baseline, 3, 6, 9, 12 and 15 months
  Differences in probing depth over the study period. PD increase must exceed a threshold of 0.8mm to be considered progression.
Mucosal recession | Baseline, 3, 6, 9, 12 and 15 months
  Measured at each of the 4 locations surrounding the implant of interest.

OTHER OUTCOMES:
Peri-implant mucosal phenotype | Baseline and 15 months
  Assessed by determining the keratinized mucosa (KM) width, measured in millimeters with a periodontal probe, at the mid-buccal aspect of the implant from the gingival margin to the mucogingival junction and the mucosal thickness, measured in millimeters, at the mid-buccal aspect of the implant, 1.5mm below the gingival margin with an endodontic spreader (0.25mm diameter) and endodontic cursor.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Ravida, DDS MS, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh School of Dental Medicine, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No